CLINICAL TRIAL: NCT01188083
Title: Effects of Dietary Fructose Reduction in Children With Hepatic Steatosis
Acronym: Sweet Bev
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Miriam Vos, MD, Principal Investigator, Emory University
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: IRB00007471; Emory-Vos-SweetBev (Other: Other)
Record Dates: First submitted 2010-06-09; First posted 2010-08-25 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Non-alcoholic Fatty-liver Disease
Keywords: NASH; non-alcoholic fatty-liver disease; Hispanic; overweight
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fructose Drink (Experimental): Subject will drink 3-8oz drinks per day for 4 weeks
  Interventions: Dietary Supplement: Fructose Drink
- Glucose Drink (Experimental): Subject will drink 3-8oz drinks per day for 4 weeks
  Interventions: Dietary Supplement: Glucose Drink

INTERVENTIONS:
Dietary Supplement: Fructose Drink — Fructose Based beverage 8 oz
  Arms: Fructose Drink
Dietary Supplement: Glucose Drink — Glucose Based beverage 8 oz per drink x 3 per day x 4 weeks
  Arms: Glucose Drink

SUMMARY:
Primary Objectives:

1. To determine whether a 4 week reduction in dietary fructose intake improves hepatic steatosis in overweight children who have a baseline high fructose consumption and hepatic steatosis.
2. To determine if a 4 week reduction of dietary fructose improves fasting plasma triglycerides, free fatty acids, very low-density lipoprotein, insulin and glucose as well as post-prandial levels in response to a high fructose meal.
3. To determine if a 4 week reduction of dietary fructose improves markers of oxidative stress.

Study Design: A blinded randomized study comparing glucose beverages to isocaloric fructose beverages administered over 4 weeks.

DETAILED DESCRIPTION:
Planned Sample Size: Phase 1) 96 subjects Phase 2) 40 subjects

Patient Population: Overweight Hispanic children with non-alcoholic fatty-liver disease age 11 to 18 years who are stable and not taking any chronic medication with no recent acute illnesses.

Definitions:

* BMI >95th %tile for age and gender
* Self-identified as Hispanic/Latino
* Baseline hepatic fat fraction > 10% (Have nonalcoholic fatty liver disease)
* Sweetened beverage intake of at least 24 ounces/day

ELIGIBILITY:
Inclusion Criteria:

* BMI > 85th %tile
* Self identified as Hispanic
* Age 11-18 years
* Baseline hepatic fat fraction >8%
* Self reported sugar beverage intake of at least 24 oz (equivalent to 3 sugar sweetened drinks per day).

Exclusion Criteria:

* Currently attempting weight gain or weight loss
* Cirrhosis visible on baseline MRI
* Renal insufficiency found on screening labs (creatinine > 2)
* Recent acute illness within past 4 weeks (defined by fever > 100.4ºF)
* Pregnancy
* Chronic illness requiring medication including diabetes
* Fasting glucose >120 on screening labs

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2009-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Hepatic Fat | 2 & 4 Weeks

SECONDARY OUTCOMES:
Plasma Triglycerides | 2 & 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Vos, Md, Principal Investigator — Emory University
Locations (1):
- Emory Children's Center, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Holzberg JR, Jin R, Le NA, Ziegler TR, Brunt EM, McClain CJ, Konomi JV, Arteel GE, Vos MB. Plasminogen Activator Inhibitor-1 Predicts Quantity of Hepatic Steatosis Independent of Insulin Resistance and Body Weight. J Pediatr Gastroenterol Nutr. 2016 Jun;62(6):819-23. doi: 10.1097/MPG.0000000000001096. PMID 26704864